CLINICAL TRIAL: NCT00664716
Title: Assessment Of Safety, Efficacy, PK&PD Of BG9924 in RA Patients Who Have Had An Inadequate Response To Conventional DMARD Therapy.
Brief Title: Assessment Of The Safety And Efficacy Of BG9924 In Rheumatoid Arthritis (RA) Participants
Acronym: RESPOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 104RA202
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; DMARD inadequate response; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Lymphotoxin-beta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): subcutaneous administration of placebo given for 12 weeks
  Interventions: Biological: Placebo
- One Dose (Experimental): BG9924 - dosage level administered as per Biogen Idec protocol
  Interventions: Biological: Baminercept alfa 1
- Second Dose (Experimental): BG9924 - dosage level administered as per Biogen Idec protocol
  Interventions: Biological: Baminercept alfa 2
- Third Dose (Experimental): BG9924 - dosage level administered as per Biogen Idec protocol
  Interventions: Biological: Baminercept alfa 3
- Fourth Dose (Experimental): BG9924 - dosage level administered as per Biogen Idec protocol
  Interventions: Biological: Baminercept alfa 4
- Fifth Dose (Experimental): BG9924 - dosage level administered as per Biogen Idec protocol
  Interventions: Biological: Baminercept alfa 5

INTERVENTIONS:
Biological: Baminercept alfa 1 — experimental - one dose level
  Other Names: BG9924; LT beta
  Arms: One Dose
Biological: Placebo — Placebo comparator
  Other Names: BG9924; LT beta
  Arms: Placebo
Biological: Baminercept alfa 2 — experimental - second dose level
  Other Names: LT beta; BG9924
  Arms: Second Dose
Biological: Baminercept alfa 3 — experimental - third dose level
  Other Names: BG9924; LT beta
  Arms: Third Dose
Biological: Baminercept alfa 4 — experimental - fourth dose level
  Other Names: BG9924; LT beta
  Arms: Fourth Dose
Biological: Baminercept alfa 5 — experimental - fifth dose level
  Other Names: LT beta; BG9924
  Arms: Fifth Dose

SUMMARY:
Safety and efficacy of BG9924 in RA participants that have had an inadequate response to disease-modifying anti-rheumatic drug (DMARD) therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of RA (functional class I - III)
* Stable dose of MTX
* Inadequate response to at least one conventional DMARD therapy

Key Exclusion Criteria:

* Serious local infection or systemic infection
* History (Hx) of recurrent infections requiring oral or parenteral anti-infective treatment
* Hx of tuberculosis (TB) or positive purified protein derivative (PPD) test during the screening period
* Clinical significant lab tests at screening
* Positive for Hep C or Hep B at screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of BG9924 in combination with methotrexate (MTX) in RA participants who have had an inadequate response to DMARD therapy | 3 months

SECONDARY OUTCOMES:
Assess the safety and tolerability of BG9924 in this participant population | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (8):
- Coordinating Research Site, San Miguel de Tucumán, Argentina
- Coordinating Research Site, São Paulo, Brazil
- Coordinating Research Site, Budapest, Hungary
- Coordinating Research Site, Cuernavaca, Mexico
- Coordinating Research Site, Torun, Poland
- Coordinating Research Site, Brăila, Romania
- Coordinating Research Site, Moscow, Russia
- Coordinating Research Site, Leeds, Yorkshire, United Kingdom

REFERENCES:
- [Derived] Bienkowska J, Allaire N, Thai A, Goyal J, Plavina T, Nirula A, Weaver M, Newman C, Petri M, Beckman E, Browning JL. Lymphotoxin-LIGHT pathway regulates the interferon signature in rheumatoid arthritis. PLoS One. 2014 Nov 18;9(11):e112545. doi: 10.1371/journal.pone.0112545. eCollection 2014. PMID 25405351